CLINICAL TRIAL: NCT07370909
Title: A Multi-center, Randomized, Double Blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of LW402 Tablets in Patients With Moderate-to-severe Atopic Dermatitis.
Brief Title: Evaluation of the Efficacy and Safety of Oral LW402 Tablets for the Treatment of Patients With Moderate-to-Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Longwood Biopharmaceuticals Co., Ltd. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LW402-III-02
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LW402 100 mg, PO BID (Experimental)
  Interventions: Drug: LW402
- LW402 150 mg, PO BID (Experimental)
  Interventions: Drug: LW402
- LW402 placebo tablets,PO.BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LW402 — LW402 tablets
  Arms: LW402 100 mg, PO BID; LW402 150 mg, PO BID
Drug: Placebo — LW402 placebo tablets
  Arms: LW402 placebo tablets,PO.BID

SUMMARY:
This Phase 3, double-blind (sponsor-open), multicenter, placebo-controlled study aims to evaluate the efficacy and safety of oral LW402 tablets in patients with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily provided informed consent and agreed to participate in the study.
* Gender: no restrictions; Age: 18 to 75 years inclusive (as of the date of signing the informed consent form).
* At screening, subjects met the Hanifin-Rajka diagnostic criteria for atopic dermatitis (AD) (Appendix 4) and had a documented AD history of ≥1 year prior to screening.
* At screening and baseline visits, subjects were required to have moderate-to-severe atopic dermatitis (AD) with all three of the following criteria satisfied:

  * Total AD lesion area ≥ 10% of body surface area (BSA)
  * Investigator's Global Assessment (IGA) score ≥ 3
  * Eczema Area and Severity Index (EASI) score ≥ 16

Exclusion Criteria:

* Subjects with a documented history of hypersensitivity to Janus kinase (JAK) inhibitors.
* Subjects with current or a history of autoimmune diseases other than atopic dermatitis (AD) (e.g., systemic lupus erythematosus [SLE], inflammatory bowel disease [IBD], Felty's syndrome, scleroderma, inflammatory myopathy, other connective tissue diseases, overlap syndrome) or other skin conditions that may interfere with AD assessment (e.g., contact dermatitis, psoriasis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving ≥75% improvement in Eczema Area and Severity Index (EASI) from baseline at Week 16 (EASI 75) | Week 16
Proportion of subjects achieving an Investigator's Global Assessment (IGA) score of 0 or 1 with a ≥2-point reduction from baseline at Week 16 | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Janzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided